CLINICAL TRIAL: NCT04689100
Title: A Phase I, Open Label, Multi-center Study to Assess the Efficacy and Safety of JMT101 in Patients With Advanced Solid Tumor.
Brief Title: Efficacy and Safety of JMT101 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-ECL
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Leucovorin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Monotherapy: Six dose levels of JMT101 will be tested according to an accelerated titration method followed by a conventional 3 + 3 study design.
  Combined with chemotherapy: Three dose levels of JMT101 will be tested by a conventional 3 + 3 study design.
  The dose-limiting toxicity (DLT) will be assessed from the first administration to the end of the first cycle (28 days).
  Interventions: Drug: JMT101
- Dose Expansion Cohort (Experimental): Once the effective dose has been determined, an expansion cohort will be opened to evaluate the efficacy and safety of the selected dose.
  Interventions: Drug: JMT101

INTERVENTIONS:
Drug: JMT101 — Monotherapy: Accelerated titration method, IV infusion QW; Conventional 3 + 3 study design, IV infusion Q2W. (28-day cycles) Combined with chemotherapy: Conventional 3 + 3 study design, IV infusion Q2W. (28-day cycles)
  Other Names: FOLFIRI(Irinotecan, Leucovorin Calcium, and Fluorouracil); mFOLFOX6((Oxaliplatin, Leucovorin Calcium, and Fluorouracil);
  Arms: Dose Escalation Cohort
Drug: JMT101 — IV infusion Q2W (28-day cycles)
  Other Names: FOLFIRI; mFOLFOX6; Irinotecan;
  Arms: Dose Expansion Cohort

SUMMARY:
This study is a Phase I, open label, multi-center study of to evaluate the safety and efficacy of JMT101 in patients with advanced solid tumor.

DETAILED DESCRIPTION:
The objective of the trial is to evaluate the safety and efficacy of JMT101 in patients with advanced solid tumor.

This study consists of two parts (Stage I and Stage II). Stage I was a dose escalation study, and Stage II was a dose expansion study.

ELIGIBILITY:
Inclusion Criteria:

* Monotherapy: Pathologically or cytologically confirmed, advanced solid tumor, harboring RAS wild type; Combined with chemotherapy: Pathologically or cytologically confirmed, locally advanced /metastatic colorectal cancer, harboring RAS and BRAF V600E wild type.
* At least 1 measurable lesion according to RECIST 1.1;
* ECOG score 0 or 1;
* Stable for more than 14 days of brain metastasis or spinal cord compression.

Exclusion Criteria:

* Receipt of any EGFR inhibitors within 5 months prior to the first dose of study treatment.
* The second primary malignant tumor was diagnosed within 5 years prior to the first dose of study treatment.
* Known hypersensitivity to any ingredient of JMT101 or their excipients;
* Major surgery within prior 4 weeks of first treatment.
* Receiving an investigational product in another clinical study within 4 weeks;
* History of serious systemic diseases;
* Pregnancy or lactating wo

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (defined by the Common Terminology Criteria for Adverse Events version 4.03 (CTCAE V4.03)). | From enrollment until 30 days after the last dose
Number of Subjects Experiencing DLTs (Dose Limiting Toxicity). | Time from the first dose of study drug up to 4 weeks
Maximum Tolerated Dose (MTD) | 28 days

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From first dose to disease progression or end of study, an average of 1 year
Disease control rate (DCR). | From first dose to disease progression or end of study, an average of 1 year
Progression free survival (PFS). | From first dose to disease progression or end of study, an average of 1 year
Overall survival (OS). | From first dose to death or end of study, an average of 1 year
Area under the concentration curve from time 0 to the concentration at last time point (AUC0-last) of JMT101. | From enrollment until 30 days after the last dose
Maximum measured plasma concentration (Cmax) of JMT101. | From enrollment until 30 days after the last dose
Time to maximum plasma concentration (Tmax) of JMT101. | From enrollment until 30 days after the last dose
Half-life (T1/2) of JMT101. | From enrollment until 30 days after the last dose
Immunogenicity profile of JMT101. | From enrollment until 30 days after the last dose
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies(ADA) and neutralizing antibodies by electrochemical luminescence(ECL).
Potential biomarkers detected in plasma or tumor issue DNA. | From enrollment up to disease progression, an average of 1 year
  The content of RAS(reticular activating system), EGFR(epidermal growth factor receptor), BRAF(B-Raf proto-oncogene) gene will be detected.

CONTACTS AND LOCATIONS:
Overall Officials: Xiugao Yang, Study Chair — Department of Medicine, CSPC Clinical Development Division
Locations (9):
- China (9):
  - Beijing Luhe Hospital. Capital Medical University, Beijing
  - Peking University Cancer Hospital, Beijing
  - The first affiliated hospital of bengbu medical college, Bengbu
  - The First People's Hospital of Changzhou, Changzhou
  - Chongqing University Cancer Hospital, Chongqing
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Zhongshan Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Henan Cancer Hospital, Zhengzhou